CLINICAL TRIAL: NCT01639456
Title: A Randomized Trial Comparing CD3/CD19 Depleted or CD3 Depleted/CD56 Selected Haploidentical Donor Natural Killer (NK) Cell Based Therapy in Older Adults With Acute Myelogenous Leukemia in First Complete Remission
Brief Title: CD3/CD19 Depleted or CD3 Depleted/CD56 Selected Haploid Donor Natural Killer Cell Treatment in Older AML in First Complete Remission
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study was abandoned and a new study was written to replace this one
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011LS151; MT2011-26 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Acute Myelogenous Leukemia
Keywords: acute myelogenous leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients Using CD3-/CD19- NK cell product (Experimental): Patients receive the apheresis product (collected day -1: enriched for NK cells using the CliniMACS® CD3 and CD19 Reagent System in combination with the large-scale tubing set (Miltenyi Biotec) to simultaneously deplete CD3+ cells to remove T-lymphocytes and deplete CD19+ cells to remove B-lymphocytes (CD3-/CD19- natural killer cells). Patients will also receive Cyclophosphamide, Fludarabine and Aldesleukin.
  Interventions: Biological: CD3-/CD19- natural killer cells; Device: CliniMACS® CD3 and CD19 Reagent System; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin
- Patients Using CD3-/CD56+ purified NK cell product (Experimental): Patients receive the apheresis product (collected day -1): purified for NK cells using the CliniMACS® CD3 Reagent System (Miltenyi Biotec) in combination with the large-scale tubing set to deplete CD3+ cells and then use the CliniMACS® CD56 Reagent System to enrich CD56+ NK cells (CD3-CD56+ natural killer cells). Patients will also receive Cyclophosphamide, Fludarabine and Aldesleukin.
  Interventions: Biological: CD3-CD56+ natural killer cells; Device: CliniMACS® CD3 and CD19 Reagent System; Device: CliniMACS® CD56 Reagent System; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin

INTERVENTIONS:
Biological: CD3-/CD19- natural killer cells — Infused on Day 0. The final CD3-/CD19- product must contain at least 20% NK cells based on previous studies using this cell product processing technique. The entire cell product will be administered except in cases where the T cell count exceeds the T cell infusion threshold. In such situations, the product volume will be adjusted to meet the lot release criteria.
  Arms: Patients Using CD3-/CD19- NK cell product
Biological: CD3-CD56+ natural killer cells — Infused on Day 0. The final CD3-/CD56+ product must contain at least 70% NK cells based on a previous study using this cell product processing technique. The entire cell product will be administered except in cases where the T cell count exceeds the T cell infusion threshold. In such situations, the product volume will be adjusted to meet the lot release criteria.
  Arms: Patients Using CD3-/CD56+ purified NK cell product
Device: CliniMACS® CD3 and CD19 Reagent System — In combination used to simultaneously deplete CD3+ cells to remove T-lymphocytes and deplete CD19+ cells to remove B-lymphocytes (CD3-/CD19-). The entire cell product will be administered except in cases where the T cell count exceeds the T cell infusion threshold. In such situations, the product volume will be adjusted to meet the lot release criteria.
Device: CliniMACS® CD56 Reagent System — CliniMACS® CD3 and CD19 Reagent System will be used in addition to CliniMACS® CD56 Reagent System to enrich CD56+ NK cells. The entire cell product will be administered except in cases where the T cell count exceeds the T cell infusion threshold. In such situations, the product volume will be adjusted to meet the lot release criteria.
  Arms: Patients Using CD3-/CD56+ purified NK cell product
Drug: Cyclophosphamide — Infused intravenously 60 mg/kg x day -5
  Other Names: Cytoxin
Drug: Fludarabine — Fludarabine 25 mg/m2 x days -6 through -2
  Other Names: Fludara
Drug: Aldesleukin — IL-2 subcutaneously at 6 million units every other day for 6 doses - begin evening of the NK cell infusion.
  Other Names: IL-2

SUMMARY:
This is a phase II trial designed to test the safety and efficacy (disease free survival [DFS]) of related donor HLA-haploidentical NK-cell based therapy for the treatment of acute myelogenous leukemia (AML). The natural killer (NK) cell product will be given to patients 60 years and older who are in a first complete remission after 1 or 2 courses of standard AML induction. After a preparative regimen of cyclophosphamide and fludarabine, patients will receive a single infusion of either CD3-/CD19- NK cells or CD3-/CD56+ NK cells followed by a short course of Interleukin-2 (IL-2) to facilitate NK cell survival and expansion.

DETAILED DESCRIPTION:
The trial will use a single-stage design and will take place in two parts. The first part will support the selection of the better NK cell product as measured by in vivo NK cell expansion. Successful in vivo NK cell expansion is defined as 40% donor DNA and 40% of lymphocytes are NK cells at day 7 post infusion OR 20% donor DNA and 20% of lymphocytes are NK cells at day 14 post infusion.

Part 1: 1:1 randomization with 10 patients per cohort to either:

1. CD3-/CD19- NK cell product or
2. CD3-/CD56+ purified NK cell product The product with better NK cell expansion will be used for the rest of the trial. If the results and safety profile are equivalent, the CD56+ selection approach will be used. If neither approach results in successful NK cell expansion, the trial will be stopped and the platform redesigned.

Part 2: complete the trial by enrolling an additional 26 patients using the product deemed successful during part 1 to estimate the primary endpoint (DFS at 12 months)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myelogenous leukemia (except acute promyelocytic leukemia) in a first complete remission (CR1) and meet the following criteria:

  * Meets the definition of complete remission by morphologic criteria including <5% blasts in a moderately cellular (> 20% cellularity) or cellular marrow.
  * Complete remission (CR) was achieved after no more than 2 cycles of standard induction chemotherapy. Early re-induction therapy based on residual disease on a day 14 bone marrow (BM) will count as a 2nd cycle. Prior therapy with demethylating agents (i.e. azacitidine) is allowed, but patients must have attained CR after standard cytotoxic therapy (defined as absolute neutrophil count (ANC) > 1000 cells/μL, platelets > 100 x 10^9/L)
  * No more than 3 months have lapsed from attainment of CR1
  * No acute myelogenous leukemia (AML) consolidation therapy administered prior to enrollment
  * Not a candidate for allogeneic stem cell transplantation
* ≥ 60 years of age
* Karnofsky performance status ≥ 70%
* Available related HLA haploidentical natural killer (NK) cell donor (sibling, offspring, or offspring of an HLA identical sibling) by at least Class I serologic typing at the A&B locus (donor age 18-75 years)
* At least 30 days since last dose of chemotherapy
* Adequate organ function within 14 days of enrollment defined as:

  * Creatinine: ≤ 2.0 mg/dL
  * Hepatic: aspartate aminotransferase (SGOT) and alanine aminotransferase (SGPT) < 5 x upper limit of institutional normal (ULN)
  * Pulmonary: oxygen saturation ≥ 90% on room air
  * Cardiac: left ventricular ejection fraction (LVEF) by echocardiogram (ECHO or MUGA) ≥ 40%, no uncontrolled angina, uncontrolled atrial or ventricular arrhythmias, or evidence of acute ischemia or active conduction system abnormalities (rate controlled a-fib is not an exclusion)
* Ability to be off prednisone and other immunosuppressive drugs for at least 3 days prior to the NK cell infusion (excluding preparative regimen pre-meds)
* Voluntary written consent

Exclusion Criteria:

* Biphenotypic acute leukemia
* New progressive pulmonary infiltrates on screening chest x-ray or chest Computed Tomography scan that has not been evaluated with bronchoscopy (when feasible). Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal, or viral infections including human immunodeficiency virus (HIV) - chronic asymptomatic viral hepatitis is allowed
* Pleural effusion large enough to be detectable on chest x-ray
* Known hypersensitivity to one or more of the study agents

Donor Selection:

* Related donor (sibling, offspring, or offspring of an HLA identical sibling) 18-75 years of age
* At least 40 kilograms
* In general good health as determined by the medical provider
* Negative for hepatitis and HIV on donor viral screen
* HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus
* Not pregnant
* Voluntary written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 1 Year
  the length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.

SECONDARY OUTCOMES:
Incidence of Infusional Toxicities | Day 100
  Patients will be monitored for adverse effects of the NK cell infusion such as rash, acute allergic reaction, bronchospasm, respiratory distress, and acute vascular leak syndrome.
Incidence of Chronic Graft-Versus-Host Disease (GVHD) | 1 Year
  Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Incidence of Acute Graft-Versus-Host Disease (GVHD) | Day 100
  Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Treatment-Related Mortality | Day 100, 1 Year and 2 Years
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Overall Survival | 1 Year and 2 Years
  The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
Disease-Free Survival | 2 Years
  the length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Miller, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri